CLINICAL TRIAL: NCT04236167
Title: Evaluating the Efficacy of an Ablative Fractional Carbon Dioxide Laser on Pathologic Symptoms in Pediatric Hypertrophic Scars: a Prospective Split-scar Controlled Trial
Brief Title: Fractional CO2 Laser Treatment of Hypertrophic Scars
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of participants to enroll. Early findings not supportive of fractionated c02 laser improving scars in population studied when used alone.
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Frankie Fraulin, Deputy Head, Department of Surgery, University of Calgary
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB17-2362
Record Dates: First submitted 2020-01-12; First posted 2020-01-22 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Cicatrix, Hypertrophic
Keywords: laser; fractional CO2 laser
MeSH Terms: conditions — Cicatrix, Hypertrophic

STUDY DESIGN:
Intervention Model Description: Prospective split scar study
Who Masked: Outcomes Assessor
Masking Description: One part of the outcomes will be assessment of clinical photographs of the scars. The assessor will be blinded to which part of the scar received the laser treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control half of scar (No Intervention): one half of the scar will receive standard scar treatment with topical products and pressure garments, but no ablative fractional CO2 laser
- Laser treatment half of scar (Experimental): The other half of the scar will receive standard scar treatment with topical products and pressure garments and, in addition, will receive ablative fractional CO2 laser treatment
  Interventions: Device: Fractional CO2 laser treatment -

INTERVENTIONS:
Device: Fractional CO2 laser treatment - — UltraPulse CO2 Laser (Lumenis, Israel). Patients will receive laser treatments at 4 to 8-week intervals for a total of 3 sessions. A combination of the SCAAR FX and Deep FX treatment modes, with or without Active FX treatment mode, will be used according to individual patient and scar characteristics. For SCAAR FX, the settings include energy (70-150mJ), density (1-5%), and frequency (150-250Hz).For Deep FX, the settings include energy (12.5-22.5mJ), density (5-15%) and frequency (300-600Hz). For Active FX, the settings include energy (80-125mJ), density (2-3%) and frequency (100-150Hz)
  Arms: Laser treatment half of scar

SUMMARY:
Executive Summary

Hypertrophic scars are irregular, raised scars that can cause debilitating symptoms including pain, pruritus, and restricted movement in nearby joints. There are also often significant psychosocial elements with these scars that are especially significant in the vulnerable pediatric population and their parents. Current scar treatment modalities are limited. In recent years, the advent of ablative fractional laser (AFL) resurfacing technology has shown great promise but there remains a need to expand high-level evidence and develop optimal laser treatment parameters for patients.

In this study, the investigators aim to evaluate the efficacy of ablative fractional CO2 laser treatment of hypertrophic scars in children and define a set of laser treatment parameters to develop a treatment protocol that maximizes the safety and efficacy of AFL therapy in the pediatric population. This will be a prospective split-scar clinical trial at Alberta Children's Hospital. A sample size of 44 scars will be sufficient to detect a clinically significant improvement in total POSAS score, our primary outcome measure. Children (age 1- 17) who present with hypertrophic scarring following an acute injury or burn may be included in the study. All patients will receive standard scar treatment modalities and will be followed by our plastic surgery team and rehabilitation team. Each scar being studied will be split into two halves which will be assigned a unique "Site ID" that will be recorded in a data collection sheet and used to identify scars for assessment. All laser treatments will be performed by a single surgeon using the UltraPulse CO2 Laser (Lumenis, Israel) and will be done at the Alberta Children's Hospital in the main operating room under a general anesthetic. Patients will receive laser treatments at 4 to 8-week intervals for a total of 3 sessions. A combination of the SCAAR FX and Deep FX treatment modes, with or without Active FX treatment mode, will be used according to individual patient and scar characteristics.

Data collection includes demographic data and original burn data. Assessment tools including the POSAS and SCAR-Q questionnaires, clinical photographs, and cutometer will be used at various time points to document changes in scar appearance and pathology over the study period. Mean values for the cutometer measurements as well as the POSAS and SCAR-Q questionnaires will be compared between laser-treated and control scar sites. Each of these datasets will be tested for normality using the Shapiro-Wilk test. Non-parametric data will be compared using Wilcoxon signed-rank test and parametric data will be compared using Student's t-tests.

DETAILED DESCRIPTION:
RATIONALE AND BACKGROUND:

Major strides in surgical care for traumatic injuries and burns over recent decades have enabled survival for wounds that would have previously been fatal. In the wake of these advancements, new challenges have emerged in managing the chronic aspects of these injuries. Among these, hypertrophic scarring remains one of our greatest unmet challenges. Hypertrophic scars are a type of pathological scar commonly formed after a traumatic injury, characterized by excessive collagen deposition during the wound-healing process that results in the appearance of an irregular, raised scar. These scars are the most common scar type formed after burn injuries with a reported incidence as high as 70%. In addition to their unpleasant appearance, hypertrophic scars can exhibit debilitating symptoms including pain, pruritus, and restricted movement in nearby joints. These symptoms often persist long after the initial wound has healed, with profound and lasting effects on patient quality of life. Stigmatization surrounding the appearance of hypertrophic scars further compounds their physical effects with psychosocial elements that are especially significant in the vulnerable pediatric population. A majority of affected children are subjected to bullying as a result of their scars and many experience increased rates of anxiety, depression, traumatic stress, and behavioral problems. Parents of affected children also experience elevated stress, depressive symptoms, and guilt. The profound, multidimensional impact of hypertrophic scarring necessitates improved treatment methods to preserve patient quality of life.

Current scar treatment modalities are limited, especially when it comes to improving the appearance of hypertrophic scars. This deficiency highlights a need to develop safe and effective new approaches that bridge the gap between conservative methods with limited efficacy and invasive measures with increased risk to patients such as surgery, laser treatment and corticosteroid injection. In recent years, the advent of ablative fractional laser (AFL) resurfacing technology has shown great promise in meeting this need with its unique combination of safety and efficacy. AFL technology fills the void between milder non-ablative lasers, which leave skin intact, and more aggressive fully ablative lasers which remove the epidermis of the entire treated surface area. While fully-ablative lasers can produce dramatic results, the large area of ablation leads to extended recovery times and increased risk of complications such as dyschromia, infection and scarring. By contrast, AFLs split the laser beam to target a dispersed pattern of the skin's surface, vaporizing precise discontinuous columns of tissue within numerous smaller areas referred to as microscopic treatment zones (MTZs). By injuring only a "fraction" of the skin, the healthy tissue surrounding the MTZs quickly regenerates and replaces the damaged tissue. Modern AFLs with ultra-pulsing technology achieve even greater efficacy by emitting the laser in rapid high-energy pulses to limit heating of adjacent tissue. By confining the treatment area to precise zones, AFLs can achieve much deeper tissue ablation than fully ablative lasers while minimizing collateral damage to surrounding tissue to maximize therapeutic effect.

Studies involving AFLs have reported a significantly diminished overall incidence of complications including those commonly associated with non-fractionated laser ablation: dyschromia, infection, and scarring. Dyschromia in the form of hyper- or hypopigmentation of the laser-treated skin is perhaps the most common side-effect that has been observed, especially in patients with darker skin types. Remarkably, using fractional ablation, the incidence of dyschromia is virtually avoided. , In addition to a reduction in overall complication rates, post-operative pain associated with AFL therapy is generally mild and well-managed even with non-opioid analgesics. General anesthesia remains the clinical consensus for avoiding intraoperative pain and thus will be implemented in this trial. Overall, AFLs are a powerful tool that can achieve a much more robust dermal remodeling response than non-ablative lasers while greatly reducing the risk of adverse effects and delayed healing seen with fully-ablative lasers and other more-invasive scar treatments.

Recent studies have examined the potential use of AFLs to treat hypertrophic scars with very promising results, documenting marked improvements in multiple aspects of scar pathology. In a large before-after cohort study, treatment of hypertrophic scars using an AFL resulted in substantial improvement of pigmentation, erythema, pliability, and thickness as measured by the gold standard Vancouver Scar Scale (VSS). The authors of this study reported a considerable reduction from 10.4 to 5.2 on the VSS within a diverse cohort of pediatric and adult patients. A more recent study that focused solely on treating pediatric burn scars with AFL also reported significant improvement with a 23% reduction in score from 89.6 to 69.2 on the Patient and Observer Scar Assessment Scale (POSAS). POSAS is similar to VSS but uniquely complements observer assessment of scars with patient-reported assessment including unprecedented assessment of pain and pruritus. The investigators will be using POSAS alongside SCAR-Q, a novel scar scale that was recently developed to provide more detailed patient-reported outcomes and unique assessment of the psychosocial impact of scars.

The demonstrated safety and efficacy of AFL resurfacing is especially attractive for application within the pediatric population. Despite promising initial reports, there remains a need to expand high-level evidence and develop optimal laser treatment parameters for patients. Existing studies rely primarily on subjective scar assessment scales for evaluating patient outcomes and few have included true objective measurements to complement their subjective data. While scar assessment scales are popular and widely accepted in both research and clinical practice, inherent subjectivity limits their reliability and significance without objective data. As such, there is a distinct need to incorporate more objective measurements into future studies. This proposed study aims to address this need by employing validated objective measurement devices in conjunction with a range of subjective measures to better evaluate the efficacy of AFLs in the treatment of pediatric hypertrophic scars. Objective measurement devices have been demonstrated to produce far better inter-rater reliability than subjective scar scales, providing essential data to more precisely examine changes in scars over the study period and substantiate subjective findings. In this study, the investigators will be using a device called a Cutometer to measure the viscoelastic properties of scars (elasticity and firmness). With more comprehensive data, our intent is to integrate and build upon recent efforts to inform further developments and facilitate the integration of AFL into the modern scar treatment paradigm.

STUDY AIM:

In this study, the investigators aim to evaluate the efficacy of ablative fractional CO2 laser treatment of hypertrophic scars in children and define a set of laser treatment parameters to develop a treatment protocol that maximizes the safety and efficacy of AFL therapy in the pediatric population.

STUDY OBJECTIVES:

1. Determine if ablative fractional CO2 laser treatment is effective in reducing pathologic symptoms and signs of hypertrophic scars including itchiness, pain, scar stiffness, and limited range of motion.
2. Determine if ablative fractional CO2 laser treatment is effective in improving the appearance of hypertrophic scars.
3. Develop a set of recommended parameters for use of ablative fractional CO2 laser treatment including timing of treatment and amount of improvement related to number of treatments.

METHODS:

Study Population The investigators propose to conduct a prospective split-scar clinical trial at Alberta Children's Hospital. A sample size of 44 scars will be sufficient to detect a clinically significant improvement in total POSAS score between the treatment and control groups of 14 points (10%) with a power of 90% and an alpha of 0.05 (Appendix). The investigators will recruit patients presenting to the outpatient burn and plastic surgery clinics at Alberta Children's Hospital over two years until reaching a sample size of 44 scars. Children (age 1- 17) who present with hypertrophic scarring following an acute injury or burn may be included in the study. To ensure the safety of participants and consistency of our data the investigators will only include patients with stable closed scars at least 3 months post wound closure. For the purposes of the study, the investigators will define wound closure as the point at which skin has been re-epithelialized and no longer requires dressings. To provide insight regarding the efficacy of early versus late laser treatment of scars, and to facilitate comparison with prior studies, the investigators will also record the age of scars being studied within two categories: scars less than 2 years post closure and scars greater than 2 years post closure. Multiple scars may be treated and studied for a single patient. Patients will be excluded from the study if they have any contraindications to general anesthesia or to receiving laser treatment such as open areas in the scar or an active infection. The investigators will also exclude patients who previously received CO2 laser therapy to the area of interest and any patients with an underlying skin disorder such as psoriasis which may influence wound healing or scar formation. Parents and patients will be consented in advance of the procedure. A document will be provided to potential participants outlining the proposal including the risks of the general anesthetic and of the laser treatment. Patients and parents will not be blinded to the treatment areas.

Study Design All patients will receive standard scar treatment modalities and will be followed by our plastic surgery team and rehabilitation team. Each scar being studied will be split into two halves which will be assigned a unique "Site ID" that will be recorded in a data collection sheet and used to identify scars for assessment. Careful initial splitting of scars should result in two regions with similar size and appearance as well as similar initial ratings on the scar scales and Cutometer measurements (described below). One half of the scar will receive standard treatment only and will be designated as the "control" area. The other half will be treated with an AFL in addition to receiving standard treatment and will be designated as the "treatment" area. The treatment area will be randomized between patients. For example, forearm scars may have the half near the elbow treated with laser in one patient but if another patient has a forearm scar, the half near the elbow in this patient may receive standard treatment only. This randomization will enable blinding of the three burn experts when reviewing the clinical photographs and help mitigate bias from scar-splitting. A transparency map will be created for each patient to map scars and measurement sites to facilitate consistency of assessments over the study period. All laser treatments will be performed by a single surgeon, Dr. Fraulin, using the UltraPulse CO2 Laser (Lumenis, Israel). Dr. Fraulin has been trained in the use of the UltraPulse CO2 laser and has used it previously in clinical practice. All laser procedures will be done at the Alberta Children's Hospital in the main operating room under a general anesthetic.

Treatment Parameters Patients will receive laser treatments at 4 to 8-week intervals for a total of 3 sessions. A combination of the SCAAR FX and Deep FX treatment modes, with or without Active FX treatment mode, will be used according to individual patient and scar characteristics. "SCAAR" stands for Synergistic Coagulation and Ablation for Advanced Resurfacing. The initial pass of the laser will be performed in the SCAAR FX treatment mode. In this mode, the laser beam penetrates skin up to a depth of 4mm to target the deeper layers of scars. For SCAAR FX, the settings include energy (70-150mJ), density (1-5%), and frequency (150-250Hz). The second pass will be done using Deep FX to treat more superficial layers of scars up to a depth of 1mm. For Deep FX, the settings include energy (12.5-22.5mJ), density (5-15%) and frequency (300-600Hz). A third mode, Active FX, is used for superficial ablation to smooth out irregular areas. It will only be used in patients with superficial irregularities in contour and dyschromia and would be used after the other two modalities as a single pass. For Active FX, the settings include energy (80-125mJ), density (2-3%) and frequency (100-150Hz).

Post-operatively patients will be instructed to take acetaminophen for pain control and to treat the laser areas with topical petroleum jelly. They will be given instructions to contact the surgeon (Dr. Fraulin) in case of any problems such as fever, increased pain, spreading redness or persistent open areas.

Data Collection and Analysis Information will be collected on each study participant including demographic data: age, sex, and Fitzpatrick skin type. Burn data will be recorded including: date of burn, anatomic location, type of burn (scald, contact, flame, flash, chemical, friction, electrical), depth of burn at treatment site and control site, time to original healing, and previous treatment of area including skin grafting.

Assessment tools including the POSAS and SCAR-Q questionnaires, clinical photographs, and Cutometer will be used at various time points to document changes in scar appearance and pathology over the study period. POSAS and Cutometer data will be collected prior to the initial treatment, just before the second treatment, and again 4-8 weeks after the last treatment. The SCAR-Q assessment and clinical photographs will only be completed at the beginning and end of the study period.

Total POSAS score will be our primary outcome for the study due to its rising prevalence in recent literature as a more reliable and comprehensive alternative to the prevailing Vancouver Scar Scale. The POSAS scar scale will be used to assess changes in scar symptoms and pathology as reported by the clinical observer and patient. POSAS will be completed twice for each scar site to independently assess both the treatment and control areas. As an additional measure, the newly-developed SCAR-Q questionnaire will be administered to provide more detailed assessment of patient-reported outcomes and unique insight regarding the psychosocial impact of scars.14 Clinical photographs of the scars will be taken before the first laser treatment and after the final laser treatment to document changes in the appearance of scars. These photographs will be reviewed by three members of the plastic surgery team with experience in burn and scar management. They will be blinded to the treatment and control areas of the scar and asked to compare and evaluate the laser-treated and control areas using photos taken at the beginning and end of the study period. Patients will not be identifiable from these photographs.

To complement the above data with objective measurements, the investigators will be using the MPA 580 Cutometer (Courage + Khazaka electronic GmbH, Germany) to assess the mechanical properties of the skin. This device applies light suction (450mbar) on a small area of the skin and measures the resulting deformation with a reflected light sensor. The exact parameters may be set by the user; however, the investigators will use consistent settings for a total measurement cycle of 4 seconds with 3 repetitions including 2 seconds of suction followed by 2 seconds for release. The Cutometer will be applied in 3 adjacent areas to record mean values for both the control and laser-treated sites of the scar as well as a separate scar-free control (either contralateral or adjacent), if available. Measurement sites will be marked on the transparency maps created for each scar to maintain the consistency of measurements. The non-invasive nature of the Cutometer and minute application pressure required means there is no pain or risk to the patient. The Cutometer software records 10 values (R0-R9) reflecting various aspects of the skin's mechanical properties. The investigators will be recording and comparing values for R0 (firmness), R1 and R2 (elasticity). Cutometer data will be recorded using the manufacturer's software (Cutometer Dual version 2.2.2.1).

Statistical Analysis:

Mean values for the Cutometer measurements as well as the POSAS and SCAR-Q questionnaires will be compared between laser-treated and control scar sites. Each of these datasets will be tested for normality using the Shapiro-Wilk test. Non-parametric data will be compared using Wilcoxon signed-rank test and parametric data will be compared using Student's t-tests. Inter-rater reliability for the assessment of the clinical photographs will be determined using intraclass correlation. Correlation between assessments will be determined using Pearson correlation. Differences will be considered statistically significant when p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Children (age 1- 17) who present with hypertrophic scarring following an acute injury or burn, with stable closed scars at least 3 months post wound closure.

Exclusion Criteria:

* Outside of age limits described above.
* Contraindications to general anesthesia.
* Open wounds in scars.
* Active infection.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change in POSAS score | Through study completion, an average of 8 months
  Unabbreviated title: Patient and Observer Scar Assessment Scale. Total minimum score = 14 maximum score = 140. Higher scores indicate worse outcome.
Change in SCAR-Q score | Through study completion, an average of 8 months
  Unabbreviated title = SCAR - Questionnaire (Patient reported outcome measure) Minimum score 29. Maximum 116. Higher score indicates worse outcome.
Change in Cutometer measurements | Through study completion, an average of 8 months
  MPA 580 Cutometer (Courage + Khazaka electronic GmbH, Germany) to assess the mechanical properties of the skin.

SECONDARY OUTCOMES:
Change in appearance on Clinical Photographs of scars | Through study completion, an average of 8 months
  Review of before and after photographs of scars by blinded observers

CONTACTS AND LOCATIONS:
Overall Officials: Frankie Fraulin, MD, Principal Investigator — Clinical Associate Professor
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Final results

REFERENCES:
- [Background] Sheridan RL. Burns. Crit Care Med. 2002 Nov;30(11 Suppl):S500-14. doi: 10.1097/00003246-200211001-00015. PMID 12528792
- [Background] Tredget EE, Levi B, Donelan MB. Biology and principles of scar management and burn reconstruction. Surg Clin North Am. 2014 Aug;94(4):793-815. doi: 10.1016/j.suc.2014.05.005. PMID 25085089
- [Background] Bombaro KM, Engrav LH, Carrougher GJ, Wiechman SA, Faucher L, Costa BA, Heimbach DM, Rivara FP, Honari S. What is the prevalence of hypertrophic scarring following burns? Burns. 2003 Jun;29(4):299-302. doi: 10.1016/s0305-4179(03)00067-6. PMID 12781605
- [Background] van Baar ME, Polinder S, Essink-Bot ML, van Loey NE, Oen IM, Dokter J, Boxma H, van Beeck EF. Quality of life after burns in childhood (5-15 years): children experience substantial problems. Burns. 2011 Sep;37(6):930-8. doi: 10.1016/j.burns.2011.05.004. Epub 2011 Jul 2. PMID 21724334
- [Background] Monstrey S, Middelkoop E, Vranckx JJ, Bassetto F, Ziegler UE, Meaume S, Teot L. Updated scar management practical guidelines: non-invasive and invasive measures. J Plast Reconstr Aesthet Surg. 2014 Aug;67(8):1017-25. doi: 10.1016/j.bjps.2014.04.011. Epub 2014 May 14. PMID 24888226
- [Background] Preissig J, Hamilton K, Markus R. Current Laser Resurfacing Technologies: A Review that Delves Beneath the Surface. Semin Plast Surg. 2012 Aug;26(3):109-16. doi: 10.1055/s-0032-1329413. PMID 23904818
- [Background] Laubach HJ, Manstein D. [Fractional photothermolysis]. Hautarzt. 2007 Mar;58(3):216-8, 220-3. doi: 10.1007/s00105-007-1286-0. German. PMID 17318467
- [Background] Metelitsa AI, Alster TS. Fractionated laser skin resurfacing treatment complications: a review. Dermatol Surg. 2010 Mar;36(3):299-306. doi: 10.1111/j.1524-4725.2009.01434.x. Epub 2010 Jan 19. PMID 20100273
- [Background] Tan KL, Kurniawati C, Gold MH. Low risk of postinflammatory hyperpigmentation in skin types 4 and 5 after treatment with fractional CO2 laser device. J Drugs Dermatol. 2008 Aug;7(8):774-7. PMID 18720695
- [Background] Wong BM, Keilman J, Zuccaro J, Kelly C, Maynes JT, Fish JS. Anesthetic Practices for Laser Rehabilitation of Pediatric Hypertrophic Burn Scars. J Burn Care Res. 2017 Jan/Feb;38(1):e36-e41. doi: 10.1097/BCR.0000000000000427. PMID 27532615
- [Background] Hultman CS, Edkins RE, Wu C, Calvert CT, Cairns BA. Prospective, before-after cohort study to assess the efficacy of laser therapy on hypertrophic burn scars. Ann Plast Surg. 2013 May;70(5):521-6. doi: 10.1097/SAP.0b013e31827eac5e. PMID 23542846
- [Background] Patel SP, Nguyen HV, Mannschreck D, Redett RJ, Puttgen KB, Stewart FD. Fractional CO2 Laser Treatment Outcomes for Pediatric Hypertrophic Burn Scars. J Burn Care Res. 2019 Jun 21;40(4):386-391. doi: 10.1093/jbcr/irz046. PMID 31225898
- [Background] Klassen AF, Ziolkowski N, Mundy LR, Miller HC, McIlvride A, DiLaura A, Fish J, Pusic AL. Development of a New Patient-reported Outcome Instrument to Evaluate Treatments for Scars: The SCAR-Q. Plast Reconstr Surg Glob Open. 2018 Apr 24;6(4):e1672. doi: 10.1097/GOX.0000000000001672. eCollection 2018 Apr. PMID 29876160
- [Background] Nedelec B, Correa JA, Rachelska G, Armour A, LaSalle L. Quantitative measurement of hypertrophic scar: interrater reliability and concurrent validity. J Burn Care Res. 2008 May-Jun;29(3):501-11. doi: 10.1097/BCR.0b013e3181710881. PMID 18388576
- [Background] Draaijers LJ, Tempelman FR, Botman YA, Tuinebreijer WE, Middelkoop E, Kreis RW, van Zuijlen PP. The patient and observer scar assessment scale: a reliable and feasible tool for scar evaluation. Plast Reconstr Surg. 2004 Jun;113(7):1960-5; discussion 1966-7. doi: 10.1097/01.prs.0000122207.28773.56. PMID 15253184
- [Background] Poetschke J, Dornseifer U, Clementoni MT, Reinholz M, Schwaiger H, Steckmeier S, Ruzicka T, Gauglitz GG. Ultrapulsed fractional ablative carbon dioxide laser treatment of hypertrophic burn scars: evaluation of an in-patient controlled, standardized treatment approach. Lasers Med Sci. 2017 Jul;32(5):1031-1040. doi: 10.1007/s10103-017-2204-z. Epub 2017 Apr 12. PMID 28401348
- [Background] Lapidoth M, Halachmi S, Cohen S, Amitai DB. Fractional CO2 laser in the treatment of facial scars in children. Lasers Med Sci. 2014 Mar;29(2):855-7. doi: 10.1007/s10103-013-1305-6. Epub 2013 Mar 26. PMID 23529372
- [Background] Miletta N, Siwy K, Hivnor C, Clark J, Shofner J, Zurakowski D, Anderson RR, Lee K, Donelan M. Fractional Ablative Laser Therapy is an Effective Treatment for Hypertrophic Burn Scars: A Prospective Study of Objective and Subjective Outcomes. Ann Surg. 2021 Dec 1;274(6):e574-e580. doi: 10.1097/SLA.0000000000003576. PMID 31469749